CLINICAL TRIAL: NCT03727607
Title: A Randomized Controlled Trial - Total Intravenous Anaesthesia Versus Inhaled Desfluran Anaesthesia in Patients Undergoing Bariatric Surgery. Postoperative Pain and Nausea
Brief Title: TIVA Versus Desfluran Anaesthesia in Patients Undergoing Bariatric Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/1659
Record Dates: First submitted 2018-03-14; First posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Total Intravenous Anesthesia; Desflurane; Obesity; Pain, Postoperative; Nausea, Postoperative
MeSH Terms: conditions — Obesity; Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Desflurane; Propofol

STUDY DESIGN:
Intervention Model Description: randomized control trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gass (Active Comparator): DESFLURANE ANESTHESIA
  Interventions: Drug: Desflurane
- TIVA (Active Comparator): TOTAL INTRAVENOUS ANESTHESIA
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Desflurane — Desflurane vs TIVA, bariatric surgery. Postoperative nausea and pain
  Other Names: PROPOFOL

SUMMARY:
Many factors during laparascopic surgery leads to PONV (postoperative nausea and vomiting), such as C02 insufflations causing peritoneal stretch and irritation and type of anaesthesia given during surgery.

The two anesthetic techniques used in bariatric surgery are gas anesthesia (Remifentanil TCI and Desfluran) and Total Intra Venous Anesthesia (TIVA) with propofol. There are studies which have shown a reduction in postoperative nausea and vomiting following TIVA, and there are publications showing no statistically significant difference.

The aim of this study was to investigate the best anaesthetic approach for obese subjects, evaluating awakening time, postoperative nausea and pain.

Our hypothesis was based on the fact that Propofol is a lipid-soluble anesthetic and therefore might have a prolonged effect in obese patients, leading to a longer awakening time along with postoperative nausea and vomiting. This hypothesis is also described earlier by obese patients have more depots (bulk fat) and also more fat surface making anaesthetics storage more easier, and also that the anesthetic will return into the circulation when the administration is stopped [18].

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥35 kg/m2 with at least one comorbid condition or BMI ≥40 kg/m2.

Exclusion Criteria:

* drug abuse
* severe mental illness
* age<18
* serious medical condition; cancer, end-stage lung disease (ASA>3) or allergies to any drugs used in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-01-30 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Awakening time after surgery | 2 hours postdose
  time noted from anaesthesia stoped to patients awake
Degree of nausea and vomiting after surgery | 48 hours postsurgery
  Noted using NRS scale (from 0-10)
Degree of pain after surgery | 48 hours post surgery
  Noted using NRS scale (from 0-10)

IPD SHARING:
Plan to Share IPD: No